CLINICAL TRIAL: NCT05748444
Title: The Relationship Between Diet and Glycemic Response and Inflammatory Markers in Children With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: büşra başpınar (Other)
Responsible Party: Sponsor-Investigator, büşra başpınar, Busra Baspinar, Ankara University
Organization: Ankara University (Other)
Other Study IDs: busrabasp92
Record Dates: First submitted 2023-01-24; First posted 2023-02-28 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis; Glucose Metabolism Disorders
Keywords: Inflammation; Cystic fibrosis; Glycemic response; Diet; Glycemic index; Blood glucose excursion; Inflammatory markers
MeSH Terms: conditions — Cystic Fibrosis; Glucose Metabolism Disorders; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cystic fibrosis: Voluntary children with cystic fibrosis aged 6-18 years with normal glucose tolerance will be included in the study.

SUMMARY:
The aim of this study is to determine the relationship between diets of children with cystic fibrosis and glycemic responses and some inflammatory markers.

DETAILED DESCRIPTION:
Cystic fibrosis is an autosomal recessive genetic disease; thick, sticky mucus accumulates in the mucin-secreting organs due to the absence or dysfunction of the cystic fibrosis transmembrane regülatör (CFTR) protein. The most commonly affected organ is the lung and the respiratory system disorder is the leading cause of death in patients with cystic fibrosis (CF). Pancreatic insufficiency is also a frequent complication in this patient group in older ages and significantly reduces life expectancy. It is argued that growth and development are adversely affected even in the stages before pancreatic insufficiency occurs. The challenges in the treatment of CFRD include dealing with increased caloric requirements for people with CF, resulting in high carbohydrate intake and frequent snacking, which exacerbates hyperglycemia. This situation causes difficulty in providing glycemic control in patients. In addition, decreased insulin secretion, as well as increased insulin resistance, delay the response to dietary glucose. This leads to an excursion of blood glucose and impaired respiratory function during the day. In addition, increased inflammation exacerbates pancreatic damage. The aim of this study is to determine the relationship between the diets of children with cystic fibrosis and glycemic responses and some inflammatory markers. In this study, general information and anthropometric measurements of patients with cystic fibrosis aged 6-18 will be recorded and their growth and development will be evaluated. With the continuous glucose monitoring system (CGMS) of the participants, the times (at least three, maximum fourteen days) when the blood glucose is below and above the target, the time in the target interval, and glucose fluctuations will be monitored. During the days of monitoring, total energy, macro-micronutrients intakes, glycemic index, and load will be calculated by asking individuals to keep a record of food consumption. The data obtained from the study will be evaluated with the SPSS package program using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* A child with cystic fibrosis between the ages of 6 and 18 who had normal glucose tolerance and volunteered to participate in the study will be included in the study.

Exclusion Criteria:

* Children with known chronic diseases such as diabetes, thyroid, liver disease (hepatitis, cirrhosis, etc.), hospitalization and/or surgery at least one month before the start of the study,
* Children who use oral/inhaled steroids, use oral antidiabetic agents, use insulin in the last month,
* Children who have had allergic bronchopulmonary aspergillosis, using intravenous or oral/inhaled antibiotic drugs at least one month ago,
* Children who wear the continuous glucose monitoring sensor for less than three days and do not keep a record of food consumption during the time it is worn

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cystic fibrosis between the ages of 6 and 18 with normal glucose tolerance will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | 90 days
  FEV1% (forced expiratory volume at one second) out of the lung function testing [ Time Frame: Within 3 months of the 7 day course of CGMS ]
Distance of shuttle walk test | 90 days
  Distance of shuttle walk test will be walked by children with cystic fibrosis. Shuttle walk test is made on floor with ten meters distance. Speed is determined according to signals from CD player.
Oral glucose tolerance test | 14 days
  The glucose values given in mmol/l after 30', 60', 90' and 120 minutes during OGTT.
Continuous glucose monitoring system (Percentage of time spent above 8mmol/l) | 14 days
  Percentage of time spent above 8mmol/l. These measurement will be gained out of the 14 day CGMS-course
Continuous glucose monitoring system (The area under the curve) | 14 days
  The area under the curve. These measurements will be gained out of the 14 day CGMS-course
Continuous glucose monitoring system (The mean glucose value (in mmol/l)) | 14 days
  The mean glucose value (in mmol/l). These measurements will be gained out of the 14 day CGMS-course
Weight in kilograms | 30 days
  Children's growth and development will be evaluated according to WHO's percentile scores.
Height in meters | 30 days
  Children's growth and development will be evaluated according to WHO's percentile scores.
Food record for three days | 3 days
  The food consumed by the children will be recorded for 3 days (on the days when the CGMS is installed).
Serum C-reactive protein (CRP) | 14 days
  Participants' serum C-reactive protein (CRP) levels will be determined.
Serum malondialdehyde (MDA) | 14 days
  Participants' serum malondialdehyde (MDA) levels will be determined.
Serum Interleukin-1-beta (IL-1B) | 14 days
  Participants' serum Interleukin-1-beta (IL-1B) levels will be determined.
Serum tumor necrosis factor-alpha (TNF-a) | 14 days
  Participants' serum tumor necrosis factor-alpha (TNF-a) levels will be determined.
Serum interleukin-6 (IL-6) | 14 days
  Participants' serum interleukin-6 (IL-6) levels will be determined.
Serum interferon-gamma | 14 days
  Participants' serum interferon-gamma levels will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of medicine, Ankara, Turkey (Türkiye)